CLINICAL TRIAL: NCT06840314
Title: VIBRENT- VIBRating vs Traditional Therapy for Treatment of ENTry Dyspareunia
Brief Title: VIBRating vs Traditional Therapy for Treatment of ENTry Dyspareunia
Acronym: VIBRENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008357
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Genito-Pelvic Pain/Penetration Disorder; Dyspareunia; Vaginismus; Pelvic Pain; Vestibulodynia; Vulvodynia (Chronic Vulvar Pain)
Keywords: genito-pelvic pain/penetration disorder; dyspareunia; entry dyspareunia; vaginismus; pelvic pain; female sexual function; pain with sex; vulvodynia; vestibulodynia
MeSH Terms: conditions — Dyspareunia; Vaginismus; Pelvic Pain; Vulvodynia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kiwi (Commercially available therapeutic vibrating pelvic floor product) (Experimental): Kiwi is a therapeutic vibrating pelvic floor product that includes an option for external massage and stimulation. The V- shaped massager, is designed to bridge anatomical variety and has three main massage ends.
  1. The cylindrical end is comparable in application to traditional vaginal dilators. However, one significant difference is its tapered shape; this allows for continuous and gradual diameter increase, as opposed to discrete increments in the traditional dilator sets. The tapered end has an optional vibration mode with 4 different intensity settings. This cylindrical shape can also be used as a tool to apply external pressure point massage to the muscles of the urogenital triangle, such as the perineal muscle and the bulbospongiosus muscles.
  2. A wider flat surface area has an additional motor to apply vibration to the glans clitoris. This end can also be used for massage.
  3. The rounded bottom end of Kiwi can be used as a broad area massage tool.
  Interventions: Device: Pelvic floor therapy
- Silicone Dilator Arm (Active Comparator): A commercially available set of graduated cylindrical vaginal dilators. The standard of care is a 6-piece, progressive-sizing, silicone dilator set. Dimensions of the silicone dilators are (WxH): (1) 0.7"x4.75", (2) 0.9"x5.25", (3) 1.0"x5.45", (4) 1.1"x5.85", (5) 1.3"x6.35", (6) 1.5"x6.85". These dilators are not battery powered, have no buttons, and no removable pieces.

INTERVENTIONS:
Device: Pelvic floor therapy — Once randomized to either the vibrating pelvic floor massage arm or the traditional vaginal dilator arm, they will receive instructions on frequency of device use and will use manufacturer's instructions for specifics of device use. We will not dictate more specific instructions on use, nor is this standard of care, as every patient is unique and will need to retain autonomy in terms of how quickly they progress in the use of the product. They will then complete a survey at 4 weeks which includes measures of sexual function and pelvic pain, as well of global impressions of improvement in their symptoms.
  Other Names: PFPT; Pelvic floor physical therapy; pelvic floor massage
  Arms: Kiwi (Commercially available therapeutic vibrating pelvic floor product)

SUMMARY:
The goal of this randomized controlled trial is to determine whether the use of a novel vibrating pelvic floor therapeutic device ("Kiwi") improves sexual function in sexually active women aged 18 and older with genito-pelvic pain and penetration disorder (GPPPD) more effectively than traditional vaginal dilators.

The main questions it aims to answer are:

1. Does the use of the Kiwi device lead to higher sexual function scores compared to traditional vaginal dilators
2. Does the Kiwi device improve sexual distress, pain, and overall symptom severity more effectively than traditional vaginal dilators?

Researchers will compare the Kiwi vibrating device to traditional cylindrical vaginal dilators to assess whether the Kiwi device results in greater improvements in sexual function and symptom relief.

Participants will:

* Be randomly assigned to use either the Kiwi device or traditional vaginal dilators.
* Use the assigned device three times per week for 15 minutes per session over four weeks.
* Complete surveys before and after the study, including assessments of sexual function, pain, and overall improvement.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) aims to evaluate the efficacy of a novel vibrating pelvic floor therapeutic device (the "Kiwi") compared to traditional vaginal dilators in improving sexual function outcomes in sexually active women aged 18 and older with genito-pelvic pain and penetration disorder (GPPPD).

The primary objective is to determine whether the Kiwi device leads to higher Female Sexual Function Index (FSFI) scores after four weeks of use compared to traditional dilators.

Secondary objectives include assessing improvements in:

* Sexual distress (Female Sexual Distress Scale - Desire/Arousal/Orgasm, FSDS-DAO)
* Pelvic pain (Vulvar Pain Assessment Questionnaire, VPAQ-screen subscale)
* Overall symptom severity (Patient Global Impression of Severity, PGI-S)
* Perceived improvement (Patient Global Impression of Improvement, PGI-I)

Participants (n=60) will be randomized into two arms:

1. Kiwi device group - a commercially available vibrating pelvic floor therapeutic product.
2. Traditional dilator group - a standard graduated cylindrical vaginal dilator set.

Participants will use their assigned device three times per week for 15 minutes per session over a four-week period. Data will be collected at baseline and at the end of the study using validated questionnaires.

The study hypothesizes that participants using the Kiwi device will demonstrate greater improvements in FSFI scores compared to those using traditional vaginal dilators, reflecting enhanced sexual function and reduced symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female at birth
* Age ≥ 18 years old
* Genito-pelvic pain/penetration disorder (per ICD-10 diagnosis codes: F52.5 Vaginismus not due to a substance or known physiological condition, F52.6 Dyspareunia not due to a substance or known physiological condition, N94.1 Dyspareunia, N94.2 Vaginismus, N94.81 Vulvodynia)

Exclusion Criteria:

* Current or prior use of a therapeutic vaginal device used to treat GPPPD
* Unmanaged genitourinary syndrome of menopause
* History of pelvic radiation
* History of genital tract malignancy
* History of female genital mutilation
* History of prior surgery for prolapse or incontinence, including vaginal mesh or midurethral sling mesh
* Silicone allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) | Four weeks
  FSFI is considered the gold standard for the measurement of sexual function in women. It's a 19-item questionnaire that uses a 5 point Likert scale ranging from 1-5, with higher scores indicating greater levels of sexual functioning on the respective item. To score the measure, the sum of each domain score is multipled by a domain factor ratio (0.6 for desire, 0.3 for arousal, 0.3 for lubrication, 0.4 for orgasm, 0.4 for satisfaction, and 0.4 for pain) in order to place all domain tools on a comparable scale. The subsequent scores are summed to derive a total FSFI score. The possible range of scores is 2-36. A score less than or equal to 26.55 reflects clinically relevant sexual dysfunction.

SECONDARY OUTCOMES:
FSDS-DAO (Female Sexual Distress Scale- Distress/Arousal/Orgasm) Questionnaire | Four weeks
  The Female Sexual Distress Scale - Distress/Arousal/Orgasm (FSDS-DAO) Questionnaire is a validated patient-reported outcome measure designed to assess sexually related distress in women, with a particular focus on distress associated with arousal and orgasmic difficulties. The FSDS-DAO consists of 15 items that assess three key domains: sexually related distress, arousal difficulties, and orgasmic dysfunction. Each item is rated on a five-point Likert scale, ranging from 0 (Never) to 4 (Always), with higher total scores indicating greater distress and dysfunction.
Primary Outcome Questionnaire (PEQ) | Four weeks
  This is a seven item questionnaire in which each question queries whether the subject has in the last four weeks attempted intercourse, insertion of one or two fingers (by self or by partner), insertion of other objects (by self or by partner). There are four responses to choose from for each question: not attempted, attempted but not successful, attempted and sometimes successful, attempted and always successful.
PGI-S- Patient Global Impression of Severity | Four weeks
  Patient Global Impression of Severity (PGI-S) is a single item questionnaire to assess a person's impression of disease severity. For purposes of this trial, it will ask participants to "Check the one number that best describes how your urinary tract condition is now" on a 4-point Likert scale ranging from (1) "normal" to (4) "severe". The PASS threshold PGI-S score is < 3.
Patient Global Impression Of Improvement (PGI-I) | Four weeks
  The Patient Global Impression of Improvement (PGI-I) is a single item questionnaire to assess an individual's impression of change in urinary symptoms. For purposes of this trial the PGI-S has been adapted by removing "taking medication" and it will ask participants to "Check the one number that best describes how your urinary tract condition is now, compared with how it was before you began this study" on a 7-point Likert scale ranging from (1) "very much better" to (7) "very much worse". The PASS threshold PGI-I score is < 3.
VPAQ-screen Subscale: Self Stimulation/Penetration Interference (Vulvar Pain Assessment Questionnaire- Screening Form) | Four weeks
  The Self Stimulation/Penetration Interference and Q7 (Vulvar Pain Assessment Questionnaire- Screening Form) asks the subject "How often do the following situations/activities cause vulvar pain?" The following situations/activities are queried: using tampons, solitary masturbation, masturbation while partner is present, solitary self penetration with fingers, solitary self penetration with sex toy.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Iglesia, MD, Principal Investigator — Medstar Washington Hospital Center National Center for Advanced Pelvic Surgery
Locations (1):
- MedStar Health, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will be collected and analyzed as an aggregate for any results.